CLINICAL TRIAL: NCT04671017
Title: A Phase I/II Randomized, Two Parts, Dose-Finding Study To Evaluate The Safety, Tolerability and Immunogenicity Of An Inactivated, Adjuvanted SARS-CoV-2 Virus Vaccine Candidate (VLA2001), Against Covid-19 In Healthy Subjects
Brief Title: Dose Finding Study to Evaluate The Safety, Tolerability and Immunogenicity of an Inactiviated, Adjuvanted SARS-CoV-2 Virus Vaccine Candidate Against Covid-19 in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VLA2001-201
Record Dates: First submitted 2020-12-15; First posted 2020-12-17 (Actual); Results first posted 2022-03-24 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: SARS-CoV-2 Virus Infection
Keywords: VLA2001; SARS-CoV-2 Virus Infection; Covid-19; inactivated-adjuvanted SARS-CoV-2 virus vaccine
MeSH Terms: conditions — COVID-19 | interventions — VLA2001 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: 1. st phase Sequential (open-label phase)
  2. nd phase Parallel Assignment (double-blinded randomized phase )
  3. rd phase Parallel Assignment (open-label phase)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 1. st phase is open-label
  2. nd phase is double-blind randomized (Participant, Investigator )
  3. rd phase is open-label phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose: VLA2001 (Experimental)
  Interventions: Biological: VLA2001
- Medium Dose: VLA2001 (Experimental)
  Interventions: Biological: VLA2001
- High Dose: VLA2001 (Experimental)
  Interventions: Biological: VLA2001
- Booster: High Dose: VLA2001 (Experimental)
  Interventions: Biological: VLA2001

INTERVENTIONS:
Biological: VLA2001 — whole virus inactivated SARS-CoV-2 vaccine adjuvanted with cytosine phospho-guanine (CpG) 1018 in combination with aluminium hydroxide

SUMMARY:
A multicenter, 3-arm randomized dose finding study in the UK to evaluate safety, tolerability and immunogenicity of a vaccine candidate against Covid-19. 150 healthy volunteers will be enrolled and receive two shots of the vaccine candidate. All participants who receive two doses of the vaccine candidate will be invited to participate in the Booster phase.

DETAILED DESCRIPTION:
The multicenter, dose finding Phase 1/2 study starts off with an open-label, dose-escalation part, thereafter, during the double-blind part of study, participants will be randomized 1:1:1 to receive the low, medium or high dose of the vaccine (VLA2001). All participants will received a total of two vaccinations intramuscularly, on day 1 and day 22.

The first 5 participants in each dose group will receive VLA2001 open label, starting with the low dose of VLA2001. If no safety concerns are identified, the next 5 subjects will receive the medium dose of the vaccine. Again, if no safety issues are identified, 5 participants will be vaccinated with the high dose of the vaccine. A Data Safety and Monitoring Board (DSMB) will review accrued safety data before randomization of the remaining 135 subjects across all sites will be initiated.

All study participants will be followed up for safety and immunogenicity up to approximately 6 months after receiving their second vaccination.

This study was extended to investigate the tolerability, safety and immungenicity of a booster vaccination with VLA2001. All study participants, in the Booster phase, will be followed up for safety and immunogenicity up to 6 months after receiving their Booster vaccination.

ELIGIBILITY:
Inclusion Criteria - Subjects who meet ALL of the following criteria are eligible for the study:

1. Participant is 18 to 55 years of age
2. Participant who has a smart phone and is willing and able to install and use the eDiary.
3. Participant has an understanding of the study and its procedures, agrees to its provisions, and voluntarily gives written informed consent prior to any study-related procedures.
4. Participant is generally healthy as determined by the Investigator
5. Participant has a Body Mass Index (BMI) of 18.0-30.0 kg/m2
6. If subject is of childbearing potential:

   1. Participant has practiced an adequate method of contraception during the 30 days before screening (Visit 0).
   2. Participant has a negative serum or urine pregnancy test at screening (Visit 0) or Visit 1, respectively.
   3. Participant agrees to employ adequate birth control measures up to Day 106 (Visit 5).

Inclusion Criteria for Booster Phase - Subjects who meet ALL of the following criteria are eligible for the Booster phase:

* B1. Participant has received complete VLA2001 primary immunization (two vaccinations according to the protocol)
* B2. Participant who has a smart phone and is willing and able to install and use the e-Diary.
* B3. Participant has an understanding of the study and its procedures, agrees to its provisions, and voluntarily gives written informed consent prior to any study-related procedures.
* B4. Participant is generally healthy as determined by the Investigator's clinical judgement
* B5. If a participant is of childbearing potential:

  1. Participant has a negative urine pregnancy test at Visit 7 prior to booster vaccination.
  2. Participant agrees to employ adequate birth control measures up to 3 months after the Booster vaccination.

Exclusion criteria - Participants who meet ANY of the following criteria are NOT eligible for this study:

1. Clinically significant infection or other acute illness, including fever ≥ 38°C within 24 hours prior to the planned study vaccination.
2. History of laboratory-confirmed SARS-CoV-2 infection.
3. Participant had close contact to persons with confirmed SARS-CoV-2 infection within 30 days prior to screening (Visit 0).
4. Participant has participated in a clinical study involving an investigational SARS-CoV-2 vaccine.
5. Participant has an acute or recent infection not due to SARS-CoV-2
6. Participant has a history of SARS-CoV-1 or MERS infection (self-reported)
7. Participant tests positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
8. Participant has received any vaccine within 30 days prior Visit 1 other than the study intervention, with the exception of the seasonal influenza vaccination.
9. Participant has abnormal findings in any required study investigations (including medical history, physical examination, and clinical laboratory) considered clinically relevant by the Investigator.
10. Participants with either medical history of or present acute or progressive, unstable or uncontrolled clinical conditions that pose a risk for participation or completion of the study, based on Investigator's clinical judgement.
11. Participants with underlying diseases with a high risk of developing severe COVID-19 symptoms if infected
12. Participant has a history of malignancy in the past 5 years other than squamous cell or basal cell skin cancer. If there has been surgical excision or treatment more than 5 years ago that is considered to have achieved a cure, the subject may be enrolled. A history of hematologic malignancy is a permanent exclusion. Participants with a history of skin cancer must not be vaccinated at the previous tumour site.
13. Participant has a known or suspected defect of the immune system, such as Participants with congenital or acquired immune deficiency
14. Participant received immuno-suppressive therapy within 4 weeks prior to Visit 1 or receipt of immunosuppressive therapy is expected during the study.
15. Participant has a history of any vaccine related contraindicating event
16. Participant presents with clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
17. Participant is pregnant, has plans to become pregnant up to Day 106 of the study or lactating at the time of enrolment.
18. Participant has donated blood, blood fractions or plasma within 4 weeks prior to Visit 1 or received blood-derived products (e.g. plasma) within 12 weeks prior to Visit 1 in this study or plans to donate blood or use blood products during the study.
19. Participant with clinically significant bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder) or prior history of significant bleeding or bruising following IM injections or venepuncture.
20. Participant has a rash, dermatological condition or tattoos that would, in the opinion of the Investigator, interfere with injection site reaction rating.
21. Participant has a known or suspected problem with alcohol or drug abuse as determined by the Investigator.
22. Participant has any condition that, in the opinion of the Investigator, may compromise the Participant's well-being, might interfere with evaluation of study endpoints, or would limit the Participant's ability to complete the study.
23. Participant is committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities).
24. Participant has participated in another clinical study involving an investigational medicinal product (IMP) or device within 4 weeks prior to Visit 0 (screening) or is scheduled to participate in another clinical study involving an IMP, or device during the course of this study.
25. Participant is a member of the team conducting the study or in a dependent relationship with one of the study team members.

Exclusion Criteria for Booster Phase - Participants who meet ANY of the following criteria are NOT eligible for Booster phase:

* B1. Clinically significant infection or other acute illness, including fever ≥ 38°C within 48 hours prior to the planned Booster vaccination.
* B2. Participant has an acute or recent infection not due to SARS-CoV-2 and is not symptom-free in the week prior to the Booster vaccination (Visit 7).
* B3. Participant has received any vaccine within 30 days prior Visit 7, with the exception of the seasonal influenza vaccination. Participants will be encouraged to receive this vaccination at least 7 days after their Booster vaccine.
* B4. Participant has abnormal findings in any required study investigations (including medical history, physical examination, and clinical laboratory) that is considered clinically relevant by the Investigator.
* B5. Participant has received immuno-suppressive therapy within 4 weeks prior to Visit 7 or is expected to receive immunosuppressive therapy during the study. Immunosuppressive therapy is defined as administration of chronic (longer than 2 weeks) prednisone or equivalent ≥ 0.05 mg/kg/day within 4 weeks prior to Visit 7 (topical and inhaled steroids are allowed), radiation therapy or immunosuppressive cytotoxic drugs or monoclonal antibodies in the previous 3 years.
* B6. Participant has clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* B7. Participant is pregnant (positive urine pregnancy test at Visit 7, respectively), has plans to become pregnant up to 3 months after the Booster vaccination.
* B8. Participant has a rash, dermatological condition that would, in the opinion of the Investigator, interfere with injection site reaction rating.
* B9. Participant has a known or suspected problem with alcohol or drug abuse as determined by the Investigator.
* B10. Participant has any condition that, in the opinion of the Investigator, may compromise the Participant's well-being, might interfere with evaluation of study endpoints, or would limit the Participant's ability to complete the study.
* B11. Participant is committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities).
* B12. Participant has participated in another clinical study involving an investigational medicinal product (IMP) or device within 4 weeks prior to Visit 7 or is scheduled to participate in another clinical study involving an IMP, or device during the course of this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valneva Clinical Development, Study Chair — Valneva Austria GmbH
Locations (4):
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - University Hospital Bristol and Weston NHS Foundation Trust, Bristol
  - Newcastle University Medical School, Newcastle
  - Southampton NIHR Clinical Research Facility, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lazarus R, Taucher C, Brown C, Corbic Ramljak I, Danon L, Dubischar K, Duncan CJA, Eder-Lingelbach S, Faust SN, Green C, Gokani K, Hochreiter R, Wright JK, Kwon D, Middleditch A, Munro APS, Naker K, Penciu F, Price D, Querton B, Riaz T, Ross-Russell A, Sanchez-Gonzalez A, Wardle H, Warren S, Finn A; Valneva Phase 1 Trial Group. Safety and immunogenicity of the inactivated whole-virus adjuvanted COVID-19 vaccine VLA2001: A randomized, dose escalation, double-blind phase 1/2 clinical trial in healthy adults. J Infect. 2022 Sep;85(3):306-317. doi: 10.1016/j.jinf.2022.06.009. Epub 2022 Jun 16. PMID 35718205

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose: VLA2001; Medium Dose: VLA2001; High Dose: VLA2001: VLA2001 whole virus inactivated SARS-CoV-2 vaccine adjuvanted with cytosine phospho-guanine (CpG) 1018 in comibinationn with aluminium hydroxide
Period: Overall Study
Arm/Group | Low Dose: VLA2001 | Medium Dose: VLA2001 | High Dose: VLA2001
Started | 51 | 51 | 51
Completed | 51 | 51 | 51
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose: VLA2001 | Medium Dose: VLA2001 | High Dose: VLA2001 | Total
Number analyzed (Participants) | 51 | 51 | 51 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (8.89) | 35.5 (9.53) | 31.3 (8.52) | 33.5 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 17 | 29 | 70
  Male | 27 | 34 | 22 | 83
Race/Ethnicity, Customized [Number; unit: count of participants]
  White | 46 | 51 | 46 | 143
  Black | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Mixed | 0 | 0 | 4 | 4
  Latin | 1 | 0 | 0 | 1
  Latin American | 2 | 0 | 0 | 2
  Latino | 1 | 0 | 0 | 1
  White European | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Solicited AEs (Local and Systemic Reactions) Within 7 Days After Any Vaccination of the Primary Vaccination Series
Time Frame: within 7 days after any vaccination
Measure: Number; unit: events
Arm/Group | Low Dose: VLA2001 | Medium Dose: VLA2001 | High Dose: VLA2001
Number analyzed (Participants) | 51 | 51 | 51
events
  Subjects with at least one Solicited Injection Site Reaction | 35 | 31 | 36
  Injection site tenderness | 32 | 23 | 34
  Injection site pain | 19 | 21 | 24
  Injection site itching | 3 | 3 | 2
  Injection site swelling | 1 | 0 | 1
  Subjects with at least one Solicited Systemic Reactions | 37 | 32 | 37
  Headache | 28 | 17 | 26
  Fatigue | 23 | 15 | 22
  Muscle pain | 18 | 15 | 17
  Nausea/Vomiting | 5 | 7 | 6
  Fever/Body temperature | 2 | 0 | 0

2. Primary Outcome: Geometric Mean Titre (GMT) for Neutralizing Antibodies Against SARS-CoV-2 Determined by Wild-type Virus Neutralizing Assay
Time Frame: Day 36
Population: Overall Number of Participants analyzed according to Per-Protocol Analysis Set. The Per-Protocol Analysis Set includes all participants who have no major protocol deviations. Participants who received an already licensed COVID-19 vaccine outside of the study or participants who received less than 2 vaccinations will be excluded.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Arm/Group | Low Dose: VLA2001 | Medium Dose: VLA2001 | High Dose: VLA2001
Number analyzed (Participants) | 51 | 49 | 50
Geometric Mean Titer | 161.1 [121.35 to 213.82] | 222.3 [171.84 to 287.67] | 530.4 [421.49 to 667.52]

3. Secondary Outcome: Frequency of Any Unsolicited AE
Time Frame: until Day 36
Measure: Number; unit: events
Arm/Group | Low Dose: VLA2001 | Medium Dose: VLA2001 | High Dose: VLA2001
Number analyzed (Participants) | 51 | 51 | 51
events
  Subjects with at least one unsolicited AE | 22 | 17 | 21
  Investigations | 10 | 8 | 8
  Red blood cell sedimentation rate increased | 5 | 4 | 5
  Aspartate aminotransferase increased | 2 | 1 | 2
  Blood bilirubin increased | 2 | 0 | 2
  Haemoglobin decreased | 0 | 0 | 2
  Lymphocyte count decreased | 0 | 1 | 1
  Red blood cells urine | 1 | 1 | 0
  White blood cell count decreased | 1 | 1 | 0
  Alanine aminotransferase increased | 0 | 0 | 1
  Blood sodium decreased | 1 | 0 | 0
  C-reactive protein increased | 1 | 0 | 0
  Neutrophil count decreased | 1 | 0 | 0
  Prothrombin time prolonged | 1 | 0 | 0
  Red blood cell count decreased | 0 | 0 | 1
  White blood cell count increased | 0 | 1 | 0
  Infections and infestations | 4 | 5 | 2
  COVID-19 | 1 | 1 | 0
  Gastroenteritis | 1 | 0 | 1
  Tooth infections | 0 | 1 | 1
  Vulvovaginal candidiasis | 0 | 2 | 0
  Epididymitis | 0 | 1 | 0
  Onychomycosis | 1 | 0 | 0
  Paronychia | 0 | 1 | 0
  Urinary tract infections | 1 | 0 | 0
  Blood and lymphatic system disorders | 4 | 2 | 4
  Neutropenia | 2 | 0 | 3
  Lymphopenia | 1 | 1 | 0
  Thrombocytopenia | 0 | 1 | 1
  Eosinophilia | 1 | 0 | 0
  Leukopenia | 1 | 0 | 0
  Microcytic anaemia | 1 | 0 | 0
  Neutrophilia | 0 | 1 | 0
  Nervous system disorders | 3 | 1 | 3
  Headache | 0 | 1 | 3
  Dizziness | 1 | 0 | 0
  Paraesthesia | 1 | 0 | 0
  Presyncope | 1 | 0 | 0
  Respiratory, thoracic and mediastinal disorders | 3 | 3 | 1
  Oropharyngeal pain | 3 | 3 | 1
  Cough | 1 | 0 | 0
  Rhinorrhoea | 0 | 1 | 0
  Sinus congestion | 1 | 0 | 0
  Injury, poisoning and procedural complications | 1 | 2 | 1
  Vaccination complications | 1 | 1 | 0
  Chillblains | 0 | 1 | 0
  Ligament sprain | 0 | 0 | 1
  Gastrointestinal disorders | 3 | 0 | 0
  Aphthous ulcer | 1 | 0 | 0
  Constipation | 1 | 0 | 0
  Diarrhoea | 1 | 0 | 0
  Gingival discomfort | 1 | 0 | 0
  General disorders and administration site conditions | 1 | 1 | 1
  Influenza like illness | 0 | 0 | 1
  Pain | 1 | 0 | 0
  Peripheral swelling | 0 | 1 | 0
  Musculoskeletal and connective tissue disorders | 1 | 2 | 0
  Arthritis | 0 | 1 | 0
  Limb discomfort | 0 | 1 | 0
  Musculoskeletal stiffness | 1 | 0 | 0
  Pain in extremity | 1 | 0 | 0
  Metabolism and nutrition disorders | 1 | 0 | 1
  Dehydration | 0 | 0 | 1
  Increased appetite | 1 | 0 | 0
  Renal and urinary disorders | 1 | 1 | 0
  Haematuria | 1 | 1 | 0
  Reproductive system and breast disorders | 1 | 0 | 1
  Dysmenorrhoea | 0 | 0 | 1
  Vaginal haemorrhage | 1 | 0 | 0
  Eye disorders | 0 | 0 | 1
  Asthenopia | 0 | 0 | 1
  Psychiatric disorders | 0 | 0 | 1
  Anxiety | 0 | 0 | 1
  Skin and subcutaneous tissue disorders | 0 | 0 | 1
  Rash erythematous | 0 | 0 | 1

4. Secondary Outcome: Frequency of Any Vaccine-related AE
Time Frame: until Day 36
Measure: Number; unit: events
Arm/Group | Low Dose: VLA2001 | Medium Dose: VLA2001 | High Dose: VLA2001
Number analyzed (Participants) | 51 | 51 | 51
events
  Subjects with at least one treatment related unsolicited AE until Day 36 | 12 | 7 | 8
  Investigations | 6 | 5 | 4
  Red blood cell sedimentation rate increased | 5 | 3 | 3
  Alanine aminotransferase increased | 0 | 0 | 1
  Blood bilirubin increased | 1 | 0 | 0
  Lymphocyte count decreased | 0 | 1 | 0
  White blood cell count decreased | 0 | 1 | 0
  Blood and lymphatic system disorders | 2 | 0 | 2
  Neutropenia | 1 | 0 | 1
  Eosinophilia | 1 | 0 | 0
  Thromocytopenia | 0 | 0 | 1
  Nervous system disorders | 2 | 0 | 1
  Dizziness | 1 | 0 | 0
  Headache | 0 | 0 | 1
  Paraesthesia | 1 | 0 | 0
  Respiratory, thoracic and mediastinial disorders | 2 | 1 | 0
  Oropharyngeal pain | 2 | 1 | 0
  Musculoskeletal and connective tissue disorders | 1 | 1 | 0
  Limb discomfort | 0 | 1 | 0
  Musculoskeletal stiffness | 1 | 0 | 0
  Gastrointestinal disorders | 1 | 0 | 0
  Diarrhoea | 1 | 0 | 0
  General disorders and administration site conditions | 1 | 0 | 0
  Pain | 1 | 0 | 0
  Infections and infestations | 0 | 0 | 1
  Gastroenteritis | 0 | 0 | 1
  Skin and subcutaneous tissue disorders | 0 | 0 | 1
  Rash erythematous | 0 | 0 | 1

5. Secondary Outcome: Frequency and Severity of Any AE
Time Frame: until Day 208
Reporting Status: Not Posted

6. Secondary Outcome: Frequency and Severity of Any Vaccine-related AE
Time Frame: until Day 208
Reporting Status: Not Posted

7. Secondary Outcome: Frequency of Any SAE
Description: All Adverse Events of Special Interest (AESIs) were treated as important medical event and were therefore be treated as SAE according to protocol.
Time Frame: until Day 36
Measure: Number; unit: events
Arm/Group | Low Dose: VLA2001 | Medium Dose: VLA2001 | High Dose: VLA2001
Number analyzed (Participants) | 51 | 51 | 51
events | 0 | 1 | 0

8. Secondary Outcome: Frequency of Any AESI
Time Frame: until Day 36
Measure: Number; unit: events
Arm/Group | Low Dose: VLA2001 | Medium Dose: VLA2001 | High Dose: VLA2001
Number analyzed (Participants) | 51 | 51 | 51
events | 0 | 1 | 0

9. Secondary Outcome: Frequency and Severity of Any SAE
Time Frame: until Day 208
Reporting Status: Not Posted

10. Secondary Outcome: Frequency and Severity of an AESI
Time Frame: until Day 208
Reporting Status: Not Posted

11. Secondary Outcome: Frequency and Severy of Solicited AEs (Local and Systemic Reactions) After the Booster Vaccination
Time Frame: until Visit 7 plus 6 days
Reporting Status: Not Posted

12. Secondary Outcome: Frequency and Severity of Any Unsolicited AE
Time Frame: until Visit 9
Reporting Status: Not Posted

13. Secondary Outcome: Frequency and Severity of Any Vaccine-related AE
Time Frame: until Visit 9
Reporting Status: Not Posted

14. Secondary Outcome: Frequency and Severity of Any SAE
Time Frame: until Visit 10
Reporting Status: Not Posted

15. Secondary Outcome: Frequency and Severity of Any AESI
Time Frame: until Visit 10
Reporting Status: Not Posted

16. Secondary Outcome: Immune Response as Measured by Neutralizing Antibody Titres Against SARS-CoV-2
Time Frame: until Day 208
Reporting Status: Not Posted

17. Secondary Outcome: Proportion of Participants With Seroconversion in Terms of Neutralizing Antibodies
Time Frame: until Day 208
Reporting Status: Not Posted

18. Secondary Outcome: Fold Increase of SARS-CoV-2 Neutralizing Antibody Titres Compared With Baseline
Time Frame: until Day 208
Reporting Status: Not Posted

19. Secondary Outcome: GMTs for IgG Antibodies Against SARS-CoV-2 Determined by ELISA
Time Frame: until Day 208
Reporting Status: Not Posted

20. Secondary Outcome: Proportion of Participants With Seroconversion in Terms of IgG Antibodies Against SARS-CoV-2, as Determined by ELISA in Participants Negative for SARS-CoV-2 at Screening
Time Frame: until Day 208
Reporting Status: Not Posted

21. Secondary Outcome: Geometric Mean Fold Rise (GMFR) From Pre-booster Time Point (Visit 7) to 2 Weeks After Booster Dose With Regards to Neutralizing Antibodies
Time Frame: until Visit 8
Reporting Status: Not Posted

22. Secondary Outcome: Geometric Mean Fold Rise (GMFR) From Pre-booster Time Point (Visit 7) to 4 Weeks After Booster Dose With Regards to Neutralizing Antibodies
Time Frame: until Visit 9
Reporting Status: Not Posted

23. Secondary Outcome: Proportion of Participants With 4-fold Increase From Pre-booster Time Point (Visit 7) to 2 Weeks After Booster Dose With Regards to Neutralizing Antibodies
Time Frame: until Visit 8
Reporting Status: Not Posted

24. Secondary Outcome: Proportion of Participants With 4-fold Increase From Pre-booster Time Point (Visit 7) to 4 Weeks After Booster Dose With Regards to Neutralizing Antibodies
Time Frame: until Visit 9
Reporting Status: Not Posted

25. Secondary Outcome: Geometric Mean Titres (GMT) Measured as Neutralizing Antibody Titres Against SARSCoV-2
Time Frame: until Visit 9
Reporting Status: Not Posted

26. Secondary Outcome: Geometric Mean Fold Rise (GMFR) From Pre-booster Time Point (Visit 7) to 2 Weeks After Booster Dose With Regards to S-protein Binding Antibodies (ELISA)
Time Frame: until Visit 8
Reporting Status: Not Posted

27. Secondary Outcome: Geometric Mean Fold Rise (GMFR) From Pre-booster Time Point (Visit 7) to 4 Weeks After Booster Dose With Regards to S-protein Binding Antibodies (ELISA)
Time Frame: until Visit 9
Reporting Status: Not Posted

28. Secondary Outcome: Proportion of Participants With 4-fold Increase From Pre-booster Time Point (Visit 7) to 2 Weeks After Booster Dose in Regards to S-protein Binding Antibodies (ELISA)
Time Frame: until Visit 8
Reporting Status: Not Posted

29. Secondary Outcome: Proportion of Participants With 4-fold Increase From Pre-booster Time Point (Visit 7) to 4 Weeks After Booster Dose in Regards to S-protein Binding Antibodies (ELISA)
Time Frame: until Visit 9
Reporting Status: Not Posted

30. Secondary Outcome: Geometric Mean Titres (GMT) Measured as IgG Antibodies Against SARS-CoV-2 (ELISA
Time Frame: until Visit 9
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the date of first vaccination until the second part of the study, where participants were followed up on Day 106 (Visit 5) and will be followed up further until Day 208/Month 7 (Visit 6), 6 months after the second vaccination.
Description: The number of participants here represent the number of healthy adults recruited in 3 dose groups (low, medium and high). Adverse event information was collected at specified time points up to the cut-off date for Day 106 (Visit 5) analysis of 30 June 2021.
Arm/Group | Low Dose: VLA2001 | Medium Dose: VLA2001 | High Dose: VLA2001
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/51 | 0/51
Other Adverse Events (participants affected / at risk) | 8/51 | 6/51 | 12/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose: VLA2001 (N=51) | Medium Dose: VLA2001 (N=51) | High Dose: VLA2001 (N=51)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose: VLA2001 (N=51) | Medium Dose: VLA2001 (N=51) | High Dose: VLA2001 (N=51)
Red blood cell sedimentation rate increased (Investigations) | 5 | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 3
Headache (Nervous system disorders) | 0 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT04671017/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT04671017/SAP_001.pdf